CLINICAL TRIAL: NCT01552811
Title: Open Study to Investigate Pancreatic Islet Mass by Positron Emission Tomography Using the Tracer [11C]5-hydroxytryptophane
Brief Title: Studies of Pancreatic Islet Mass by Positron Emission Tomography (PET)
Status: Completed | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Per-Ola Carlsson, Professor, Uppsala University Hospital
Other Study IDs: AS Dnr2011/439
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Type 1 diabetes
- healthy controls

SUMMARY:
This study investigates the hypothesis that differences in beta-cell mass in patients with diabetes and healthy individuals can be monitored by the positron emission tomography (PET) tracer [11C]5-hydroxytryptophane.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with type 1 diabetes
* Adult, healthy controls

Exclusion Criteria:

* Pregnancy
* Impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult, type 1 diabetic patients Healthy controls
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Difference in pancreatic uptake of % injected dose (ID) [11]5-hydroxy tryptophan between healthy volunteers and patients with long-standing type 1 diabetes | To be measured at Positron emission tomography investigation for all study persons.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Eriksson O, Espes D, Selvaraju RK, Jansson E, Antoni G, Sorensen J, Lubberink M, Biglarnia AR, Eriksson JW, Sundin A, Ahlstrom H, Eriksson B, Johansson L, Carlsson PO, Korsgren O. Positron emission tomography ligand [11C]5-hydroxy-tryptophan can be used as a surrogate marker for the human endocrine pancreas. Diabetes. 2014 Oct;63(10):3428-37. doi: 10.2337/db13-1877. Epub 2014 May 21. PMID 24848067